CLINICAL TRIAL: NCT00902252
Title: Multi-National Phase III Vitala™ 12-Hour Wear Test
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Dheerendra Kommala, MD / VP of Clinical Development, Convatec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-0196-08-A720
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual/Natura®/Vitala™ (Experimental): All subjects will wear usual product for 21 days, followed by Natura® for 14 days and followed by Vitala™ for 159 days.
  Interventions: Device: Usual; Device: Natura®; Device: Vitala™

INTERVENTIONS:
Device: Usual — All subjects will wear their usual pouching system for the first 21 days of the study.
Device: Natura® — All subjects will wear the Natura® Flexible Skin Barrier with Flange (Stomahesive® or Durahesive®) in the US and Natura® Stomahesive® Flexible Skin Barrier with Flange in Europe for 14 days.
Device: Vitala™ — After the successful completion of Stages 1 and 2, subjects will enter the "ramp up" schedule to allow the subject to adjust to the device. This consists of weekly increases in wear time of the Vitala™ device beginning with 4 hours of daily wear per week (Days 36 to 42), followed by 6 hours of daily wear time per week (Day 43 to 49), followed by 8 hours of daily wear time (Days 50 to 56) and progressing to 12 hours of daily wear per week (Day 57 to 215).

SUMMARY:
The purpose of this clinical study is to demonstrate that the Vitala™ Continence Control Device is both safe and effective when worn up to 12 hours per day.

ELIGIBILITY:
Inclusion Criteria:

* Is of legal consenting age.
* Is able to read, write, and understand the study, the required procedures, and the study related documentation.
* Has signed the informed consent.
* Has an end colostomy of at least 12 weeks duration with formed or semi- formed effluent.
* Is able to wear a Natura® skin barrier wafer flange in size 45mm or 57 mm.
* Is willing to remove and replace the skin barrier wafer after three days, more often if desired.
* Has a stoma that protrudes no more than 2 cm at rest.
* Has demonstrated success in wearing a traditional pouching system. (Investigator judgment)
* Is willing to participate in the trial for a total of 215 days. (approximately 7 months)
* Is willing to meet with the investigator for a total of 12 scheduled visits plus additional visits as deemed necessary by the investigator.
* Has the ability to do complete self-care.

Exclusion Criteria:

* Has known skin sensitivity to any component of the products being tested.
* Has a skin rating of "2" or greater according to the Skin Rating Scale.
* Is receiving radiation in the area of the pouching system.
* Is receiving chemotherapy other than a stable regimen of maintenance chemotherapy.
* Requires a pouch belt while wearing Vitala
* Requires convexity or a moldable skin barrier.
* Has participated in a clinical study within the past 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety | 159 Days
  Will be assessed by measuring the frequency of adverse events relating to the stoma (including gastrointestinal, stomal and surrounding skin events), microbiology profile and stomal vascularity.
Restoration of Continence | 159 days
  Absence of fecal leakage around the device.

SECONDARY OUTCOMES:
Efficacy | 215 Days
  Will be assessed by the following: measurement of health economic outcomes, resource use, security, wear time, comfort, control of odor, control of noise, ease of use during application and removal, subject acceptance of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Dheerendra Kommala, MD, Study Director — ConvaTec Inc.
Locations (12):
- United States (8):
  - Private Practice, Tuscon, Arizona
  - ET Nursing Services, Jacksonville, Florida
  - Washington County Hospital, Hagerstown, Maryland
  - Restored Images, Kansas City, Missouri
  - Image Specialties, Saint Joseph, Missouri
  - Mt. Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Colon and Rectal Surgery, Reynoldsburg, Ohio
- Germany (2):
  - University Hospital Freiburg, Freiburg im Breisgau
  - Private Practice, Triwalk
- United Kingdom (2):
  - Homerton University Hospital NHS, London
  - Chelsea and Westminster Hospital, London